CLINICAL TRIAL: NCT06867289
Title: Study of the Efficacy of Moderate Sedation With Intra-NAsal Dexmedetomidine Monitored by EEG MOnitoring
Acronym: DINAMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-02-CHRMT
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Procedural Sedation and Analgesia; Pediatric ALL
Keywords: MRI; dexmedetomidine; EEG
MeSH Terms: conditions — Agnosia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: A cohort of patients with an indication for DEX sedation for brain NMRI will be included. EEG monitoring will be performed in addition to usual practice, prior to DEX administration and for 20 minutes prior to NMRI, to enable calculation of the PSI sedation score (at 0, 10, 20 minutes). Sedation will also be assessed by the PSSS clinical score at 0, 10, 20 minutes after DEX administration, as well as at 150 minutes after DEX.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG Monitoring and PSSS clinical score (Experimental): All participants receive an EEG monitoring.
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — EEG monitoring will be performed in addition to the usual practice, before DEX administration and for 20 minutes before NMRI, to enable calculation of the PSI sedation score (at 0, 10, 20 minutes). Sedation will also be assessed by the PSSS clinical score at 0, 10, 20 minutes after DEX administration, as well as at 150 minutes after DEX.

SUMMARY:
This is a prospective, monocentric diagnostic study aiming to evaluate whether a sedation score obtained by a per-procedural electroencephalogram (EEG), the PSI score, could identify patients for whom a 2 μg/kg dose of DEX would not be sufficient for the successful performance of cerebral NMRI, and who could therefore benefit from a higher dosage of DEX (4 μg/kg).

DETAILED DESCRIPTION:
For some children, brain MRI is a particularly important examination for etiological assessment or for monitoring the progress of neurological diseases. It can sometimes be complicated to perform, due to the age and/or pathology of the child concerned. Impossibility, postponement or the need for a general anaesthetic are constraints that should be avoided as far as possible. Procedural sedation with dexmedetomidine (DEX) can be administered intra-nasally. This technique offers good results and safety of use. Nevertheless, the failure rate is 20% to 30%, and may depend on the dosage of DEX used (indicated doses vary from 2 to 4 μg/kg). This study aims to evaluate whether a sedation score obtained by a per-procedural electroencephalogram (EEG), the PSI score, could identify patients for whom a 2 μg/kg dose of DEX would not be sufficient for the successful performance of cerebral NMRI, and who could therefore benefit from a higher dosage of DEX (4 μg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Indication of DEX sedation for brain NMRI at the CHR de Metz-Thionville

  * in a patient aged between 12 months and 5 years or
  * for a patient aged between 5 and 18 whose cooperation during the examination appears compromised (previous failure, autism spectrum disorders, etc.).
* Membership of a social security scheme
* Free and informed consent obtained from the patient's legal guardian(s).

Exclusion Criteria:

* Weight < 10 kg
* Patients with contraindications to the use of DEX

  * Hypersensitivity to the active ingredient or to any of the excipients listed in the section on "Hypersensitivity".
  * Advanced heart block (level 2 or 3), unless pacemaker implanted
  * Uncontrolled hypotension
  * Acute cerebrovascular pathologies
* Patients with nasal obstruction
* Parental refusal of DEX administration
* Minors under guardianship
* Minors under judicial sanction

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Prediction of complete NMRI success | 20 minutes after DEX administration
  To describe the predictive value (ROC curve) of the PSI score assessed 20 minutes after administration of 2 μg/kg of DEX intranasally, for complete success in performing brain NMRI in children under 5 years of age, or over 5 years of age with risk of failure.
  Successful NMRI is defined as:
  * Complete if all prescribed sequences can be interpreted without reservation,
  * Partial if some of the sequences cannot be interpreted or are subject to reservations by the radiologist,
  * Absent if the examination is cancelled or if all sequences are uninterpretable or subject to reservations.
  PSI score: evaluated on EEG, the score varies from 0 to 100.

SECONDARY OUTCOMES:
Complete or partial success in performing brain NMRI in children under 5 years of age, or over 5 years of age with risk of failure. | 20 minutes after DEX administration
  Area under the ROC curve for prediction of complete or partial success of NMRI according to PSI score.
  Successful NMRI is defined as:
  * Complete if all prescribed sequences can be interpreted without reservation,
  * Partial if some of the sequences cannot be interpreted or are subject to reservations by the radiologist,
  * Absent if the examination is cancelled or if all sequences are uninterpretable or subject to reservations.
Predictive value (ROC curve) of the PSI score for successful completion of brain MRI in children under 5 years of age, or over 5 years of age with risk of failure. | 20 min after DEX administration
  Area under the ROC curve for prediction of complete success of NMRI according to PSI score by patient age under or over 5 years old
  Successful NMRI is defined as:
  * Complete if all prescribed sequences can be interpreted without reservation,
  * Partial if some of the sequences cannot be interpreted or are subject to reservations by the radiologist,
  * Absent if the examination is cancelled or if all sequences are uninterpretable or subject to reservations.
  PSI score: evaluated on EEG, the score varies from 0 to 100.
Predictive value (ROC curve) of the PSSS score for successful completion of brain MRI in children under 5 years of age, or over 5 years of age with risk of failure. | 20 min after DEX administration
  Area under the ROC curve for prediction of complete or partial success of NMRI according to PSSS score at 20 minutes
  Successful NMRI is defined as:
  * Complete if all prescribed sequences can be interpreted without reservation,
  * Partial if some of the sequences cannot be interpreted or are subject to reservations by the radiologist,
  * Absent if the examination is cancelled or if all sequences are uninterpretable or subject to reservations.
  PSSS score: ranges from 0 (deepest sedation) to 5 (shallowest sedation) depending on the observation of clinical signs in children
Correlation between PSI and PSSS scores | at 0, 10, 20 and 150 minutes after DEX administration
  Describe the correlation between PSI score and PSSS score PSI scores at 0, 10, 20 and 150 minutes after DEX administration and PSSS scores at 0, 10, 20 and 150 minutes after DEX administration
Complications (Quality of recovery) | at 150 minutes after DEX administration
  PSSS score: ranges from 0 (deepest sedation) to 5 (shallowest sedation) depending on the observation of clinical signs in children
Complications (Blood Pressure) | at 0, 10, 20 and 150 minutes after DEX administration
  mmHg
Complications (Heart Rate) | at 0, 10, 20 and 150 minutes after DEX administration
  bpm
Complications (Oxygen Saturation) | at 0, 10, 20 and 150 minutes after DEX administration
  SaO2 (%)
Complications (allergic reactions) | at 0, 10, 20 and 150 minutes after DEX administration
  number and types

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Charlotte CULLIER, MD, Principal Investigator — CHR Metz Thionville Hopital Femme Mère Enfant
Locations (1):
- CHR Metz-Thionville Hopital Femme-Mère Enfant, Metz, France